CLINICAL TRIAL: NCT01732861
Title: A MULTICENTER, PHASE 1B, OPEN-LABEL STUDY TO DETERMINE THE SAFETY AND ACTIVITY OF CC-292 IN COMBINATION WITH LENALIDOMIDE IN SUBJECTS WITH RELAPSED AND/OR REFRACTORY CHRONIC LYMPHOCYTIC LEUKEMIA / SMALL LYMPHOCYTIC LYMPHOMA
Brief Title: Safety Study of CC-292 and Lenalidomide in Subjects With Chronic Lymphocytic Leukemia/ Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-292-CLL-001; 2012-003766-41 (EudraCT Number)
Record Dates: First submitted 2012-11-14; First posted 2012-11-26 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Leukemia Lymphocytic Chronic B-Cell
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — spebrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-292 + Lenalidomide (Experimental)
  Interventions: Drug: CC-292; Drug: Lenalidomide

INTERVENTIONS:
Drug: CC-292 — CC-292-will be given twice daily on Days 8-28 of Cycle 1 and on Days 1-28 of the remaining 28-day cycles.
Drug: Lenalidomide — Lenalidomde will be given once daily on Days 1-28 of 28-day cycles.

SUMMARY:
This is a dose finding study using a 3 + 3 dose escalation and expansion design to determine a Not Tolerated Dose (NTD), Optimal Biological Effect Dose (OBE) and / or Maximum Tolerated Dose (MTD). These data will be used to establish a Recommended Phase 2 Dose (RP2D) for the combination of CC-292 and lenalidomide in subjects with Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
This dose finding study uses a 3 + 3 dose escalation and expansion design to establish the recommended Phase 2 dose. The starting dose is CC-292 375 mg twice daily and Lenalidomide 10 mg once daily. After review of the data for dose limiting toxicities (DLTs), the second dose level will be enrolled. Doses for this second cohort are CC-292 500 mg twice daily and lenalidomide 10 mg once daily. Additional doses of lenalidomide in combination with CC-292 may be evaluated to accurately determine the maximum tolerated dose. Once the maximum tolerated dose and/or optimal biologic effect has been ascertained, an expansion cohort of 24 subjects may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age and older at the time of signing the informed consent document (ICD).
* Body weight at least 50 kg.
* Must have a documented diagnosis of CLL/SLL (International Workshop on Chronic Lymphocytic Leukemia IWCLL Guidelines - Hallek 2008) by investigator assessment.
* Have failed at least 1 previous treatments for CLL/SLL, and have relapsed and/or refractory disease following last prior treatment defined as CLL/SLL that does not achieve at least a partial response (PR) to therapy or that progresses within 6 months of treatment.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 2 or less.
* Life expectancy of at least 3 months from time of signing ICD.
* Females of childbearing potential (FCBP) must have a negative medically supervised pregnancy test prior to starting study therapy and agree to ongoing pregnancy testing during and after end of study therapy; commit to continued abstinence from heterosexual intercourse or agree to use, comply with two effective methods of contraception without interruption, 28 days prior to starting study drug, during study therapy, and for 28 days after discontinuation of study therapy.
* Male subjects must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy, throughout study drug therapy and dose interruption, and for 28 days after end of study therapy; agree to not donate semen or sperm during study drug therapy and for 28 days after end of study drug therapy.
* All subjects must understand that lenalidomide could have a potential teratogenic risk, agree to abstain from donating blood with taking lenalidomide therapy and following discontinuation of study drug therapy; have an echocardiogram (ECG) or multigated acquisition (MUGA) scan of the heart demonstrating left ventricular ejection fraction (LVEF) at least 50% or the institution's lower limit of normal; have recovered from adverse, toxic effects of prior therapies to equal to or less than 1 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.03 except for alopecia and peripheral neuropathy.

Exclusion Criteria:

- Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.

* Autologous stem cell transplant within 3 months prior to the time of signature on the ICD Informed Consent Document.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring parenteral antibiotics; uncontrolled diabetes mellitus; chronic symptomatic congestive heart failure; unstable angina pectoris, angioplasty, stenting, or myocardial infarctions within 6 months prior to the time of signature on the ICD; clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia. Subjects with controlled atrial fibrillation that is asymptomatic are eligible.
* Pregnant or lactating females.
* Prior history of malignancies, unless the subject has been free of the disease for 5 years or more prior to the time of signature on the ICD. Exceptions to the 5 years or more time limit include history of basal cell carcinoma of the skin; squamous cell carcinoma of the skin; carcinoma in situ of the cervix; carcinoma in situ of the breast; carcinoma in situ of the bladder; incidental histologic finding of prostate cancer (Tumor/Nodes/Metastasis [TNM] stage of T1a or T1b).
* Known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV).
* Known seropositivity for hepatitis C virus (HCV); hepatitis B virus (HBV).
* Subjects who are at a high risk for a thromboembolic event and are not willing/able to take venous thromboembolic event (VTE) prophylaxis.
* Any of the following laboratory abnormalities:

  1. Absolute Neutrophil Count (ANC) ≤ 1,000 cells/mm3 (1.0 x 109/L)
  2. Platelet count ≤ 50,000/mm3 (50 x 109/L) unless secondary to bone marrow involvement by recent bone marrow aspiration and bone marrow biopsy
  3. Serum Aspartate Transaminase/Serum Glutamic-Oxaloacetic Transaminase (AST/SGOT) or Alanine Transaminase/Serum Glutamic-Pyruvic Transaminase (ALT/SGPT) > 3.0 x upper limit of normal (ULN) or > 5.0 x ULN in cases of documented liver involvement
  4. Serum bilirubin > 1.5 x ULN or > 3.0 x ULN in cases of Gilbert's Syndrome and documented liver involvement by lymphoma;
  5. Calculated creatinine clearance using the Cockcroft-Gault formula (Cockcroft,1976)
  6. Corrected QT interval (QTc) prolongation (defined as a QTc > 450 msec for males and > 470 msec for females [Fridericia's correction]) or other clinically significant ECG abnormalities as assessed by the investigator.
* Chemotherapy, radiotherapy, investigational anticancer therapy or major surgery within 28 days of Day 1 dosing.
* Use of systemic corticosteroids in doses greater than prednisone equivalent to 20 mg/day within 3 weeks prior to study drug dosing.
* Concomitant use of medicines known to cause QT prolongation or torsades de pointes.
* Chronic use of H2 antagonists or proton pump inhibitors or their use within 7 days of first dose.
* Gastrointestinal abnormalities including the inability to take oral medication, requiring intravenous alimentation, or prior surgical procedure affecting absorption.
* Prior treatment with Btk (Bruton's tyrosine kinase) inhibitors.
* Any live vaccinations within 3 weeks from first dose.
* History of hypersensitivity to immunomodulatory drugs (IMiDs) (eg, lenalidomide, thalidomide, pomalidomide).
* Disease transformation (ie, Richter's Syndrome [lymphomas] or prolymphocytic leukemia).
* Patients with uncontrolled hyper or hypothyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12-28 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 5 years
  Number of participants with adverse events

SECONDARY OUTCOMES:
Percentage of Participants Who Have Received Some Form of Response | Up to 2 years
  Response rate is defined as the percentage of participants who have achieved some form of response including: a Complete Response (CR), a CR with incomplete bone marrow recovery, a Nodular Partial Response (PR), a Nodal PR or a PR with lymphoctyosis) based on the International Workshop for Chronic Lymphocytic Leukemia and lymphoma guidelines (IWCLL).
PK-Cmax | Up to 15 days
  Maximum observed plasma concentration
PK-Tmax | Up to 15 days
  Time to maximum observed plasma concentration
PK-λz | Up to 15 days
  Terminal phase rate constant, determined by linear regression of the terminal points of the log-linear plasma concentration-time curve. Visual assessment will be used to identify the terminal linear phase of the concentration
PK-t1/2 | Up to 15 days
  Estimate of the terminal elimination half-life in plasma
PK-AUC (0-t) | Up to 15 days
  Area under the plasma concentration-time curve from time zero to time t, where t is the last measurable time point
PK-AUC0-∞ | Up to 15 days
  Area under the plasma concentration time curve from time zero extrapolated to infinity.

CONTACTS AND LOCATIONS:
Overall Officials: David Liu, MD, Study Director — Celgene
Locations (11):
- United States (6):
  - Clearview Cancer Institute Oncology Specialties, P.C, Huntsville, Alabama
  - Horizon Oncology Center, Lafayette, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - The West Clinic, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Austria (5):
  - Universitatsklinik fur Innere Medizin, Innsbruck
  - AKh Linz, Linz
  - Universitatsklinik der PMU, Salzburg
  - Allgemeines Krankenhaus Wien, Vienna
  - Medizinische Abteilung-Zentrum fur Onkologie und Hamatologie, Vienna